CLINICAL TRIAL: NCT04657159
Title: Health-economic Evaluation of Interventional Pain Management Compared to Pain Rehabilitation
Status: Completed | Type: Observational
Sponsor: Eques Indolor AB (Other)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: IPM-PRP2020
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2010-2016: Patients treated 2010-2016
  Interventions: Other: Pain rehabilitation program
- 2017-2019: Patients treated 2017-2019
  Interventions: Other: Pain rehabilitation program

INTERVENTIONS:
Other: Pain rehabilitation program — Effect on health related quality of life och health-care consumption after rehabilitation

SUMMARY:
The overall aim of the study is to evaluate interventional pain management. This is done in three steps:

1. To find matched controls to the patients in the study on cost-effectiveness of IPM and compare the results.
2. To calculate cost-effectiveness of PRP during the period 2010-2016, on a national level.
3. To calculate cost-effectiveness of PRP during the period 2017-2019, after the changed guidelines for PRP in Sweden.

The two last steps are to provide a background to the results of IPM, and to see if the results in the subgroup of matched controls of PRP-patients differ from the results from the whole population.

DETAILED DESCRIPTION:
Chronic pain is one of the major health problems globally, according to the WHO 'global burden of disease' studies. Previously, the investigators have performed a study on a feasible approach to be able to treat zygapophyseal joint pain in the thoracic region, similar to the established methods for treatment in the lumbar and cervical regions which have been published. The study showed that there was a significant improvement in health related quality of life (HRQoL) after treatment, and that there were no difference in the results depending on if it was the cervical, thoracic or lumbar region that was treated. The study had ethical approval (Dnr 2012-446-31M) and is registered here at clinicaltrials.gov.

Another study explored the health economic aspects of interventional pain management (IPM). The investigators aimed to do this in comparison with pain rehabilitation programs, and therefore further ethical approval was searched and gained (2012-446-31M, 2017-542-32, 2018- 507-32) An health-economic evaluation of only IPM was performed showing that patients after treatment of diagnosed pain-focuses in zygapophyseal joint pain not only improve their HRQoL but they also reduce their medication, reduced their health-care consumption and gained in ability to work. The cost per quality adjusted life years gained was below the threshold for cost-effective health-care according to the threshold-levels defined by the national Board of Health and Welfare in Sweden. But the investigators need a larger population to select from in order to get matched controls among patients that have been through pain rehabilitation programs.

This study therefore aims to explore the national register of pain rehabilitation both in order to find matched controls and in order to make a cost-effectiveness study of pain rehabilitation program as it is performed in Sweden.

ELIGIBILITY:
Inclusion Criteria:

Been through pain rehabilitation program

Exclusion Criteria:

-

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have been treated with pain rehabilitation programs and that have been registered prospectively in the national register for pain rehabilitation in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 15611 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 1 year
  EQ-5D index

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lindholm, Study Director — PhD
Locations (2):
- Sweden (2):
  - Department of Epidemiology and Global Health Umeå University, Umeå
  - Smärtkliniken Eques Indolor, Vallentuna

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is restricted by law in Sweden and any sharing needs a specific approval from ethics board